CLINICAL TRIAL: NCT04490863
Title: Noninvasive Hemoglobin Spot Check Repeatability and Reproducibility in a Blood Donation Setting
Brief Title: Noninvasive Hemoglobin Repeatability and Reproducibility in a Blood Donation Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SDBB0005
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Results first posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Healthy; Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test subjects (Experimental): All subjects are enrolled and receive Rad-67 Pulse oximeter & DCI Mini sensor for measurement of hemoglobin.
  Interventions: Device: Rad-67 Pulse oximeter & DCI Mini sensor

INTERVENTIONS:
Device: Rad-67 Pulse oximeter & DCI Mini sensor — Noninvasive pulse oximeter that measures hemoglobin

SUMMARY:
The primary objective of this clinical investigation is to report on the repeatability and reproducibility of SpHb measurements from Rad-67 devices and DCI Mini sensors used to screen prospective blood donors at a donation center.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Weight at least 110 pounds
* Subjects with the intention of being screened for eligibility to donate blood
* The subject has given written informed consent to participate in the study

Exclusion Criteria:

* Subjects with skin abnormalities at the planned application sites that may interfere with sensor application, per directions-for-use (DFU) or trans-illumination of the site, such as burns, scar tissue, infections, abnormalities, etc.
* Subjects unwilling to remove nail polish or acrylic nails
* Subjects with blood cancers such as leukemia
* Subjects with hemoglobin disorders such as sickle-cell anemia and thalassemia or with known history of infectious diseases such as HIV/AIDS, syphilis, hepatitis, etc.
* Subjects with self-disclosed/known pregnancy at the time of enrollment
* Subjects deemed not suitable for the study at the discretion of the investigator
* Subjects unlikely to be able to refrain from excessive motion during data collection. Excessive motion includes postural changes, making hand gestures, involuntary muscular movements, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Blood Bank - Site 1, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Subjects
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Test Subjects
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 23
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2
  Race: Native Hawaiian or Other Pacific Islander | 1
  Race: Black or African American | 1
  Race: White | 12
  Race: More Than One Race | 1
  Race: Unknown or Not Reported | 1
  Race: Mexican | 7
  Race: Middle Eastern | 1
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Coefficient of Variation of Rad-67
Description: Coefficient of variation will be computed using Repeatability and Reproducibility variance.
Time Frame: Approximately 90 minutes per subject
Measure: Number; unit: Coefficient of Variation percentage
Arm/Group | Test Subjects
Number analyzed (Participants) | 26
Coefficient of Variation percentage | 4.50

ADVERSE EVENTS:
Time Frame: Approximately 90 minutes per subject
Arm/Group | Test Subjects
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT04490863/Prot_SAP_000.pdf